CLINICAL TRIAL: NCT04681365
Title: A Phase I Study of an 'In-house' Developed Prototype Powered Air Purifying Respirator (PAPR) for Use as Personal Protective Equipment (PPE) for Healthcare Workers (Bubble PAPR)
Brief Title: Evaluating Bubble-PAPR for Healthcare Workers
Acronym: BubblePAPR
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: B00991
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Simulation Suite: Participating staff will use BubblePAPR and evaluate its function in the non-clinical simulation suite, ensuring that simulated tasks appropriate to role can be undertaken safely whilst wearing the Bubble
  Interventions: Other: Staff will wear and evaluate Bubble-PAPR (non-CE marked PAPR)
- Low-Risk Clinical Environment: Participating staff will use BubblePAPR and evaluate its function in the usual clinical environments (wards, ICUs or Emergency Departments) but with patients who are considered low risk (ie non-COVID-19).
  Interventions: Other: Staff will wear and evaluate Bubble-PAPR (non-CE marked PAPR)
- High-Risk Clinical Environment: Participating staff will use BubblePAPR and evaluate its function in the usual clinical environments (wards, ICUs or Emergency Departments) but with patients who are considered high risk (ie suspected or confirmed COVID-19).
  Interventions: Other: Staff will wear and evaluate Bubble-PAPR (non-CE marked PAPR)

INTERVENTIONS:
Other: Staff will wear and evaluate Bubble-PAPR (non-CE marked PAPR) — Staff will wear and evaluate the Bubble PAPR instead of usual PPE consisting of FFP3/N95 facemasks. This novel, non-CE marked prototype PPE is a Powered air Purifying Respirator and is used 'in house' (not approved for use outside of the Sponsor organisation)

SUMMARY:
This project will produce a low cost, ergonomic, hood integrated PAPR for use initially within the NHS. It will focus on user centred design, engineering optimisation, feasibility testing, certification and intellectual property protection.

This study will evaluate the pre-CE marked Bubble PAPR prototype PPE in the clinical environment and gather usability data from consenting participants (staff).

DETAILED DESCRIPTION:
Aim: To develop low cost, ergonomic, personal protective equipment to prevent virus transmission to NHS healthcare workers.

This project aims to address these problems by taking a user centred design approach to develop and manufacture a highly functional Hood Integrated Personal Air Purifying Respirator (HI-PAPR) at a low cost. The design team brings together Manchester University NHS Foundation Trust (MFT) ICU frontline clinical staff, an experienced product design consultancy, Designing Science Limited (DSL) and the technical expertise of the School of Engineering at the University of Manchester (UoM). The project will run through a rapid design and evaluation cycle in simulated and clinical environments to refine the concept to meet regulatory requirements. The final product could be used in primary/secondary care and in the community and will be ready for wide-scale manufacture and supply for the UK NHS within six months of the project start.

This study will evaluate Bubble PAPR in the clinical environment and gather usability data from frontline healthcare staff.

We hypothesise that:

* The Bubble PAPR will meet or exceed the British and European standards for PAPRs.
* That participating staff who subsequently use the PAPR will rate the PPE as:
* More comfortable than current PPE
* Safer than current PPE
* Easier to communicate with colleagues than current PPE
* Easier to communicate with patients than current PPE

Our research question is:

• Do clinical staff report that the Bubble PAPR is more comfortable than current FFP3 facemasks.

ELIGIBILITY:
Inclusion Criteria:

Provision of informed consent; bedside clinical staff (medical, nursing, allied healthcare professional) who manage patients with COVID-19 disease during routine clinical duties.

Exclusion Criteria:

Refusal to participate; unable to, or unwilling to wear the Bubble PAPR

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All individuals will be considered for inclusion in this study regardless of age, disability, gender reassignment, marriage and civil partnership, pregnancy and maternity, race, religion and belief, sex, and sexual orientation except where the study inclusion and exclusion criteria EXPLICITLY state otherwise.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is that participating staff rate Bubble PAPR to be more comfortable than current PPE. | 1month
  Primary outcome measure is 'Comfort' as defined by Q17 of the questionnaire ("Please indicate how comfortable the Bubble PAPR is") on a 7-point Likert scale bounded by 1 (very uncomfortable) through to 7 (very comfortable).

SECONDARY OUTCOMES:
Staff rate Bubble PAPR as safer than current PPE | 1month
Staff rate Bubble PAPR as easier to communicate with colleagues than existing PPE | 1month
Staff rate Bubble PAPR as easier to communicate with patients than existing PPE | 1month

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McGrath BA, Shelton CL, Gardner A, Coleman R, Lynch J, Alexander PG, Cooper G. Bubble-PAPR: a phase 1 clinical evaluation of the comfort and perception of a prototype powered air-purifying respirator for use by healthcare workers in an acute hospital setting. BMJ Open. 2023 May 8;13(5):e066524. doi: 10.1136/bmjopen-2022-066524. PMID 37156585